CLINICAL TRIAL: NCT05075018
Title: Evaluation of Musculoskeletal Problems, Endurance, Quality of Life and Physical Activity Level in Healthcare Professionals With COVID-19 Infection and Without COVID-19 Infection
Brief Title: Musculoskeletal Problems and Endurance in Healthcare Professionals With and Without COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Other Study IDs: AIBU-FTR-ETY-02
Record Dates: First submitted 2021-09-28; First posted 2021-10-12 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Respiratory Infection
Keywords: COVID-19; Muscle Endurance; Musculoskeletal Problems; Healthcare Workers
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare Workers with COVID-19 Infection: Healthcare workers who have been diagnosed with COVID-19 in the past and currently do not have COVID-19 disease constitute this group
  Interventions: Other: Observational
- Healthcare Workers without COVID-19 Infection: Healthcare workers who have not been diagnosed with COVID-19 in the past and currently do not have COVID-19 disease constitute this group
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Individuals' musculoskeletal problems will be evaluated with the Cornell Musculoskeletal Disorder Questionnaire, quality of life, physical activity, Nottingham Health Profile physical activity International Physical Activity Questionnaire, endurance stabilizer device, functional exercise capacity 1 minute sit and stand test, shortness of breath using the Modified Borg Scale. Measurements will be made only once.

SUMMARY:
The effects of frequency and severity of physical complaints and symptoms on general well-being, sleep and quality of life are known. However, in the COVID-19 process, the disease has very different effects, both physical and psychological, and some symptoms persist even if the disease is overcome; In addition to these, the fact that the measures taken throughout the country prompt individuals to take measures to protect themselves from the disease and make it compulsory under some conditions intertwine many different dimensions of the disease on human health and significantly affect daily life. In this context, our first aim in this study is to compare factors such as musculoskeletal problems, physical activity level, endurance and quality of life in healthcare workers with and without COVID-19. Seconder aim is to examine the relationships between factors such as musculoskeletal problems, physical activity level, endurance and quality of life, and to examine the effect levels of the parameters by performing regression analyzes depending on the result.

DETAILED DESCRIPTION:
COVID-19 (The coronavirus disease 2019), COVID-19 infection with a wide variety of symptoms such as pain, shortness of breath, high fever, loss of taste and smell, diarrhea and can even progress to a very serious condition such as acute respiratory distress syndrome. It is a common disease that has manifested itself worldwide in the last 1 year as a disease and was declared a pandemic by the World Health Organization on March 11, 2020.

80% of the cases have mild or asymptomatic disease, and 20% need treatment in hospital conditions. Although the disease affects different age groups, it generally affects people aged 60 and over more. It can take weeks to get over the disease; however, some symptoms persist even after the infection has cleared. The continuation of physical, cognitive and psychological problems in COVID-19 patients recovering from the acute phase of the disease is called 'Post-COVID-19 Syndrome'. Symptoms of the disease include fever, dry cough and shortness of breath, as well as common musculoskeletal problems such as muscle pain, joint pain and fatigue, anxiety, depression, poor sleep quality and decreased quality of life, and difficulties in daily living activities. Moreover, the course and prevalence of the disease and its severity in our country as well as in the world have developed a new psychological pressure about the disease and revealed the situation of coronavirus phobia, and even this affects the mood and sleep quality of individuals. It has been shown that depression and anxiety are observed, especially in patients with severe respiratory-related symptoms, both during the active period of the disease and during the period when the symptoms continue despite the recovery of the disease, and the quality of life is adversely affected.

The effects of frequency and severity of physical complaints and symptoms on general well-being, sleep and quality of life are known. However, in the COVID-19 process, the disease has very different effects, both physical and psychological, and some symptoms persist even if the disease is overcome; In addition to these, the fact that the measures taken throughout the country prompt individuals to take measures to protect themselves from the disease and make it compulsory under some conditions intertwine many different dimensions of the disease on human health and significantly affect daily life. In this context, our first aim in this study is to compare factors such as musculoskeletal problems, physical activity level, endurance and quality of life in healthcare workers with and without COVID-19. Seconder aim is to examine the relationships between factors such as musculoskeletal problems, physical activity level, endurance and quality of life, and to examine the effect levels of the parameters by performing regression analyzes depending on the result.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering,
* Being a healthcare worker

Exclusion Criteria:

* Using psychiatric medication
* No surgery in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are health workers working in a health institution; It will consist of two groups, those who have been diagnosed with COVID-19 in the past and those who have not been diagnosed with COVID-19 in the past.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of the Endurance | 15 minutes
  Endurance of deep cervical flexor muscles and core muscles (Transversus abdominous muscle and lumbar multifidus muscle) will be evaluated with The Stabilizer Pressure Biofeedback Unit. The device will be placed on the measured muscles; Individuals will be asked to maintain their position at the desired pressures. It will give the individual the time to maintain the desired value and the pressure score. High scores indicate that endurance is preserved; low scores reflect loss of endurance.

SECONDARY OUTCOMES:
Cornell Musculoskeletal Discomfort Questionnaire | 5 minutes
  The scale divides the body into 20 distinct regions. Each region's score ranges from 0 to 90. It is understood that the higher the score, the greater the pain, the severity of the pain and the limitation of the pain.
Nottingham Health Profile | 10 minutes
  The Nottingham Health Profile will be used to assess health-related quality of life. The questionnaire consists of 38 items and consists of six subsections related to health status: Energy, pain, emotional reactions, sleep, social isolation and physical activity. Each section is scored between 0-100. 0 indicates best health, 100 indicates worst health.
International Physical Activity Questionnaire | 5 minutes
  Physical activity level will be measured with the International Physical Activity Questionnaire. The questionnaire evaluates parameters such as vigorous activities, moderate activities, walking and sitting activities. The higher the score, the higher the physical activity; A low score indicates physical inactivity.
1 minute sit to stand test | 2 minutes
  Sit and stand test can be performed to evaluate functional exercise capacity, lower extremity muscle strength and endurance. Individuals are asked to cross their arms over their shoulders and sit and stand up for 30 seconds as fast and as long as they can, and the number of sit-ups is recorded. High scores indicate good functional capacity, strength and endurance; low scores indicate functional impairment.
Modified Borg Scale | 2 minutes
  Dyspnea assessment will be made with the Modified Borg Scale. Scoring ranges from 0 to 10 points. High scores indicate high dyspnea; low scores indicate low breathlessness.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem TÜTÜN YÜMİN, Assoc. Prof., Study Director — Bolu Abant İzzet Baysal University
Locations (1):
- Düzce Atatürk Devlet Hastanesi, Düzce, Turkey (Türkiye)